CLINICAL TRIAL: NCT04451278
Title: RESting-state Functional MRI for Prediction of Post-surgical Prognosis In Pediatric Drug-Resistant Epilepsy
Acronym: RESPIRE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-A01561-38
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resting-state functional MRI (r-fMRI): The MRI examination will be performed on a 3T multi-parametric MRI. Compared to the standard protocol, patients will benefit from an additional fMRI-r sequence, called resting state, and performed before injection of gadoline contrast.
  A neuropsychological evaluation is performed as part of the 6 months prior to the procedure. These data will be used as a basis for the evaluation of language visual and language recovery.

SUMMARY:
Resting-state functional MRI (r-fMRI) has emerged in recent years to analyze resting networks. It allows, without active participation of the patients, to identify and analyze the different functional brain networks. The analysis of r-fMRI can be done thanks to the graph theory, which is based on the based on the calculation of quantifiable parameters applied to the functional network studied, making it possible to assess its effectiveness.

To the knowledge of the investigators, no study has used graph theory applied to r-fMRI data in order to obtain parameters useful for the useful parameters for the individual prognosis of children who have to be operation for drug-resistant lesional epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 6 and 18 years
* Receiving an MRI for lesional drug-resistant epilepsy
* Affiliated or beneficiary of a social security plan
* Whose parents or guardians have received information about the study and have given their express consent to participate in the study

Exclusion Criteria:

* Contraindication to absolute or relative MRI (in particular, pregnant or breastfeeding women)
* History of intracranial surgery
* MRI performed under general anesthesia

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from 6 to 18 years old receiving an MRI as part of a preoperative assessment of lesion epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Determine the prognostic value of topological parameters measured on local r-fMRI on the surgical success at one year of patients operated for drug-resistant epilepsy. | One year
  The variables measured with functional MRI will correspond to topological parameters of functional connectivity measured locally at the level of the lesion: the degree, the clustering coefficient and path length. Surgical success will be evaluated by a score of 1 on the modified Engel classification at one year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sidney KRYSTAL, Principal Investigator — Adolphe de Rothschild Fondation Hospital
Locations (1):
- Fondation A De Rothschild, Paris, PARIS, France

IPD SHARING:
Plan to Share IPD: No